CLINICAL TRIAL: NCT02794181
Title: Study of Zika Virus and Related Arbovirus Infections in Deferred Blood Donors
Brief Title: Zika Virus and Related Arbovirus Infections in Deferred Blood Donors (ZVADD)
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 160124; 16-CC-0124
Record Dates: First submitted 2016-06-08; First posted 2016-06-09 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03-14

CONDITIONS: Zika Virus; Dengue Virus; Chikungunya Virus Infections
Keywords: Transfusion-Transmitted Infections; Dengue Virus; Chikungunya Virus; Natural History; Blood Transfusion
MeSH Terms: conditions — Zika Virus Infection; Chikungunya Fever; Transfusion Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

Zika virus is mostly passed on by the bite of an infected mosquito. It usually causes mild illness. But in pregnant women it can cause serious birth defects to the baby. The virus can also spread by blood transfusion and sexual intercourse. This is why the U.S. Food & Drug Administration (FDA) recommended that people should not give blood if possibly exposed to Zika virus. Dengue virus and chikungunya virus are passed by the same mosquitoes as Zika virus. These can cause severe reactions if passed through transfused blood.

Donated blood is usually not tested for these three viruses. Researchers want to count the infections in people who have been exposed because of travel or sexual exposure. They want to learn the risk these viruses might pose to the U.S. blood supply. They also want to study the natural history of these viruses by following infected people over time.

Objective:

To study the risk of Zika, dengue, and chikungunya viruses to the U.S. blood supply.

Eligibility:

Adults age 18 or older who were turned down for donating blood because of possible exposure to certain viruses.

Design:

Participants will have blood and urine tests. They will answer questions about their travel.

They will be called in about a week with virus test results.

Participants with negative results do not have any more study visits.

Participants with positive results will be asked to stay in the study for 6 months. They will have weekly clinic visits and tests until results are negative for 2 straight weeks. Once test results are negative, they will have monthly visits. Visits will include physical exams, blood and urine samples, and optional semen samples from men.

Most people will have 3-4 weekly visits and 5 monthly visits.

DETAILED DESCRIPTION:
Zika virus (ZIKV) is an Aedes species mosquito-transmitted Flavivirus responsible for an ongoing epidemic in over twenty countries and territories in the Caribbean, and in North, Central and South America. A 20-fold increased risk of microcephaly has been reported in newborns of infected mothers in Brazil. Of nine identified pregnant travelers returning to the U.S. from areas with local ZIKV infection, five have experienced severe neonatal outcomes.

ZIKV can be transmitted via blood transfusion and by sexual exposure to a ZIKV-infected man. In response, AABB (formerly the American Association of Blood Banks) made recommendations and the Food and Drug Administration (FDA) issued guidance for donor deferral based on 1) travel to locations with active ZIKV transmission; or for 2) sexual exposure to a man who has traveled to an area with active ZIKV transmission. Further, Aedes species mosquito vectors that transmit ZIKV also transmit dengue virus (DENV) and chikungunya virus (CHIKV). Areas with local ZIKV transmission also commonly have local DENV and CHIKV transmission. DENV and CHIKV are transmissible via blood transfusion and can result in severe outcomes in transfusion recipients.

The primary aims of this study are to: 1) assess the prevalence of ZIKV, DENV and CHIKV infection (RNA-positives) among adults who attempted to donate blood but were deferred because of travel to places with local transmission of ZIKV, DENV and/or CHIKV (travel-deferred donors); 2) assess the prevalence of ZIKV infection (RNA-positives) among adults who attempted to donate blood who were deferred due to potential sexual exposure to ZIKV infection; 3) assess the prevalence of ZIKV, DENV and CHIKV infection (RNA-positives) among blood donors whose blood or platelets were collected and who called back to report any illness within 2 weeks of donation; and to 4) study the 24-week natural history of ZIKV, DENV and CHIKV infection among deferred adult donors who tested RNA-positive for any of these agents.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults who traveled within the past month to places with local transmission of ZIKV, DENV and/or CHIKV who would otherwise be eligible to donate blood;
* Volunteer adult blood donors or potential blood donors who are deferred from blood donation because they tested positive for Zika virus.
* Volunteer adult blood and platelet donors (blood donors) who present to the NIH Clinical Center Department of Transfusion Medicine (DTM) and the Fishers Lane Donor Center are eligible for study enrollment if they:

  1. Are deferred because of travel to an area with active ZIKV transmission within the past 4 weeks; or
  2. Are deferred because of sexual contact during the past 4 weeks with a sexual partner who traveled to an area with active ZIKV transmission in the 3 months prior to that instance of sexual contact; or
  3. Are deferred because of travel to a malaria-endemic area; and returned from the area in the past month; or
  4. Have donated blood or platelets AND within 2 weeks of donation they called the NIH DTM or Fishers Lane Donor Centers to report any signs or symptoms of infection, AND they traveled to an area with active transmission of ZIKV, DENV or CHIKV within the past 4 weeks (from symptom onset); OR had sexual contact within the past 4 weeks (from symptom onset) with a sexual partner who traveled to an area with active ZIKV transmission in the 3 months prior to that instance of sexual contact.

EXCLUSION CRITERIA:

Potential donors who do not meet the inclusion criteria are excluded. Potential donors under 18 years of age, paid or research blood donors and pregnant women are excluded from enrollment. Children are not eligible to donate blood without parental consent and the frequency of number of follow-up visits places an undue burden on school age children. Paid or research blood donors are not representative of the normal blood donor population. Pregnant women are not eligible to donate blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06-08; Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of ZIKV, DENV and CHIKV infection (RNA-positives) among travel-deferred adult blood donors in the study population. | Time 0; among RNA-positives: weeks 1,2,3,4,5,6,7,8,9,10,11,12,16,20,24
Prevalence of ZIKV infection (RNApositives) among adult blood donors with a history of potential sexual exposure to ZIKV infection, in the study population. | Time 0; among RNA-positives: weeks 1,2,3,4,5,6,7,8,9,10,11,12,16,20,24
24-week Natural History of ZIKV, DENV and CHIKV (RNA-positives). | weeks 1,2,3,4,5,6,7,8,9,10,11,12,16,20,24

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Allison, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Musso D, Nhan T, Robin E, Roche C, Bierlaire D, Zisou K, Shan Yan A, Cao-Lormeau VM, Broult J. Potential for Zika virus transmission through blood transfusion demonstrated during an outbreak in French Polynesia, November 2013 to February 2014. Euro Surveill. 2014 Apr 10;19(14):20761. doi: 10.2807/1560-7917.es2014.19.14.20761. PMID 24739982
- [Background] Alter HJ, Stramer SL, Dodd RY. Emerging infectious diseases that threaten the blood supply. Semin Hematol. 2007 Jan;44(1):32-41. doi: 10.1053/j.seminhematol.2006.09.016. PMID 17198845
- [Background] Lanciotti RS, Kosoy OL, Laven JJ, Velez JO, Lambert AJ, Johnson AJ, Stanfield SM, Duffy MR. Genetic and serologic properties of Zika virus associated with an epidemic, Yap State, Micronesia, 2007. Emerg Infect Dis. 2008 Aug;14(8):1232-9. doi: 10.3201/eid1408.080287. PMID 18680646